CLINICAL TRIAL: NCT01294631
Title: An Open-Label, Two-Period, Fixed-Sequence Study to Explore the Effects of Multiple Doses of Hydrochlorothiazide on the Pharmacodynamics, Pharmacokinetics, and Safety of Multiple Doses of Canagliflozin in Healthy Subjects
Brief Title: A Pharmacodynamics, Pharmacokinetics, and Safety Study of Hydrochlorothiazide and Canagliflozin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017851; 28431754DIA1034
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: Canagliflozin; JNJ-28431754; Hydrochlorothiazide; Pharmacokinetic; Pharmacodynamic
MeSH Terms: interventions — Canagliflozin; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): Canagliflozin 300 mg once daily and HCTZ 25 mg once daily Period 1: canagliflozin tablets oral 300 mg once daily on Days 1 to 7 followed 14 days later by Period 2.
  Period 2: HCTZ tablets oral 25 mg once daily for Days 1 to 28 followed by canagliflozin tablets oral 300 mg once daily taken with HCTZ tablets oral 25 mg once daily on Days 29 to 35..
  Interventions: Drug: Canagliflozin 300 mg once daily and HCTZ 25 mg once daily

INTERVENTIONS:
Drug: Canagliflozin 300 mg once daily and HCTZ 25 mg once daily — Period 1: canagliflozin tablets, oral, 300 mg, once daily on Days 1 to 7 followed 14 days later by Period 2.
  Period 2: HCTZ tablets, oral, 25 mg, once daily for Days 1 to 28 followed by canagliflozin tablets, oral, 300 mg, once daily taken with HCTZ tablets, oral 25 mg, once daily on Days 29 to 35..

SUMMARY:
The purpose of the study is to evaluate the effects of multiple doses of hydrochlorothiazide and canagliflozin on the concentrations of each drug in the blood and the concentration of glucose in the blood and urine in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a single-center, open-label study with 2 study periods where volunteers and study staff will know the names and doses of assigned study treatments. All volunteers will receive the same treatment. Canagliflozin (a sodium-glucose cotransporter 2-inhibitor) is currently under development to lower blood sugar levels in patients with Type 2 diabetes mellitus (T2DM), and hydrochlorothiazide (HCTZ) is a drug indicated for the treatment of patients with mild to moderate hypertension. During Period 1, volunteers will take canagliflozin 300 mg once daily for 7 days (Days 1 to 7) and during Period 2, volunteers will take HCTZ 25 mg once daily for 28 days (Days 1 to 28), and then starting on Day 29, will take canagliflozin 300 mg once daily and HCTZ 25 mg once daily for 7 days (Days 29 to 35). Period 1 and Period 2 will be separated by a minimum of 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index (BMI, a measure of a person's weight in relation to height) between 18 and 30 kg/m2, inclusive, and a body weight of not less than 50 kg

Exclusion Criteria:

* History of or current clinically significant medical illness as determined by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose
* Known allergy to canagliflozin or any of the excipients of the formulation of canagliflozin

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Urine glucose concentration | At protocol-specified time points up to Day 36 in Period 2

SECONDARY OUTCOMES:
Plasma concentration of canagliflozin | Up to Day 36 in Period 2
Plasma concentration of hydrochlorothiazide (HCTZ) | Up to Day 36 in Period 2
Plasma glucose concentration | At protocol-specified time points up to Day 36 in Period 2
Blood pressure and heart rate measurements | Up to Day 46 in Period 2
Plasma and urine electrolyte assessment | Up to Day 36 in Period 2
The number and type of adverse events reported | Up to Day 46 in Period 2

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Devineni D, Vaccaro N, Polidori D, Rusch S, Wajs E. Effects of hydrochlorothiazide on the pharmacokinetics, pharmacodynamics, and tolerability of canagliflozin, a sodium glucose co-transporter 2 inhibitor, in healthy participants. Clin Ther. 2014 May;36(5):698-710. doi: 10.1016/j.clinthera.2014.02.022. Epub 2014 Apr 13. PMID 24726680